CLINICAL TRIAL: NCT01073501
Title: Efficacy of Pregabalin in the Management of Chronic Uremic Pruritus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Shavit Linda MD, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111.CT.IL
Record Dates: First submitted 2010-02-17; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Uremic Pruritus
Keywords: UREMIC PRURITUS; PREGABALIN; UP
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Placebo versus pregabalin
  Interventions: Drug: Placebo
- Pregabalin (Experimental): Placebo versus pregabalin
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 25 mg (Lyrica; Pfizer, Germany) or placebo will be administered orally daily at the end of hemodialysis sessions in dialysis patients or every evening in non dialysis CKD patients. The dose will be increased up to 50 mg if no improvement of pruritus will be established at the end of first week of the study
  Arms: Pregabalin
Drug: Placebo — Pregabalin 25 mg (Lyrica; Pfizer, Germany) or placebo will be administered orally daily at the end of hemodialysis sessions in dialysis patients or every evening in non dialysis CKD patients. The dose will be increased up to 50 mg if no improvement of pruritus will be established at the end of first week of the study
  Arms: Placebo

SUMMARY:
Uraemic pruritus (UP) remains a frequent and distressing problem in patients with advanced or end-stage renal disease. Its intensity ranges from sporadic discomfort to complete restlessness during both the day- and night-time and its distribution varies significantly over time. Many attempts have been made to relieve this bothersome symptom in affected patients, however with generally limited success. Incidence of UP varies widely between studies and seems to decline over the last 30 years (from 85% in the 1970s and 50-60% in the 1980s to a 22% in the 2000s) (Gunal AI).

We use Pregabalin for the relief of diabetic neuropathic pain in patients on haemodialysis in our centre. In addition to neuropathic pain, several of our patients have complained of pruritus and after Pregabalin treatment, their pruritus has promptly and completely resolved. Accordingly, we intend to conduct a double-blind, placebo-controlled, crossover trial to assess the effectiveness of Pregabalin in chronic UP.

ELIGIBILITY:
Inclusion Criteria:

1. History of pruritus of >8 weeks duration.
2. Severity of pruritus of 7 or more defined by visual analogue scale.
3. No improvement by oral antihistamines or skin moisturizers.
4. Discontinuation of any medication with presumed antipruritic effects at least 1 week before the study.
5. Negative pregnancy test result for all participating women of childbearing age;

Exclusion Criteria:

1. Known allergy to Pregabalin
2. Any acute illness;
3. Liver cirrhosis
4. Active dermatological disorder other than UP
5. Decompensated heart failure;
6. Inability to give informed consent;
7. Poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Reduction of UP by more than 50% after Pregabalin administration | 2012

SECONDARY OUTCOMES:
Reduction of chronic pain of various origin and improvement in insomnia after Pregabalin administration | 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264